CLINICAL TRIAL: NCT04847986
Title: A Guided Eight-week Online Acceptance and Commitment Therapy (ACT) Intervention for Distressed Family Caregivers of People With Dementia: A Mixed-methods Pilot Study
Brief Title: Guided Eight-week Online Acceptance and Commitment Therapy for Distressed Family Caregivers of People With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Occupational Therapy Foundation (Other)
Responsible Party: Principal Investigator, Areum Han, Assistant professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AOTFIRG21Han
Record Dates: First submitted 2021-04-08; First posted 2021-04-19 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Psychological Distress
Keywords: Acceptance and Commitment Therapy; Alzheimer's Disease; Burden; Caregivers; Dementia; Mindfulness; Psychological health; Quality of life; Self-compassion; Stress; Depression; Anxiety; Guilt; Grief
MeSH Terms: conditions — Alzheimer Disease; Dementia; Psychological Well-Being; Depression; Anxiety Disorders | interventions — Acceptance and Commitment Therapy; Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acceptance and commitment therapy (ACT) group (Experimental): 8 weekly ACT sessions individually guided by a trained coach through Zoom videoconferencing with psychoeducation materials provided
  Interventions: Behavioral: acceptance and commitment therapy (ACT)
- Control group (Sham Comparator): care as usual with psychoeducation materials provided
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: acceptance and commitment therapy (ACT) — Caregivers assigned to this intervention group will receive individual ACT sessions guided by a trained coach for one hour per week over 8 weeks through Zoom videoconferencing with psychoeducation materials provided.
  Arms: acceptance and commitment therapy (ACT) group
Behavioral: Control group — The control group will receive care as usual with psychoeducation materials provided.
  Arms: Control group

SUMMARY:
The pilot randomized controlled trial aims to assess effects of a guided online acceptance and commitment therapy (ACT) intervention on distressed family caregivers of people with dementia (PwD) compared to the control group. A total of 24 family caregivers of PwD who meet the inclusion criteria will be recruited and randomized to either the intervention or control group. Exploratory hypotheses are that the ACT group will show decreases in caregivers' psychological distress and burden and improvements in QoL and engagement in meaningful activities at posttest and 1-month follow-up, compared to the control group. Also, the project will evaluate the feasibility of recruitment, adherence, and retention of caregivers and explore caregivers' experiences in the ACT intervention through semi-structured interviews at posttest. As part of the pretest, we will also explore caregivers' perceived impacts of COVID-19 on daily lives.

DETAILED DESCRIPTION:
The pilot randomized controlled trial aims to assess effects of a guided online acceptance and commitment therapy (ACT) intervention on distressed family caregivers of people with dementia (PwD) compared to the control group. A total of 24 family caregivers of PwD who meet the inclusion criteria will be recruited and randomized to either the intervention or control group. Caregivers assigned to the intervention group will receive individual ACT sessions guided by a trained coach for one hour per week over 8 weeks through Zoom videoconferencing with supplemental psychoeducation materials provided. Caregivers assigned to the control group will receive care as usual with psychoeducation materials provided. Outcomes regarding caregivers' mental health will be collected at three time points (i.e., pretest, posttest, and 1-month follow-up) and compared between groups over time. Exploratory hypotheses are that the ACT group will show decreases in caregivers' psychological distress and burden and improvements in QoL and engagement in meaningful activities at posttest and 1-month follow-up, compared to the control group. Also, the project will evaluate the feasibility of recruitment, adherence, and retention of caregivers and explore caregivers' experiences in the ACT intervention through semi-structured interviews at posttest. As part of the pretest, we will also explore caregivers' perceived impacts of COVID-19 on daily lives.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling adults (age 18 or over) who are currently taking the primary responsibility for the care of a relative with dementia living in the community
* devoting at least four hours daily to the care of the relative with dementia
* having at least mild symptoms of psychological distress as measured by the Depression, Anxiety and Stress Scale (DASS-21; Antony et al., 1988)
* having a computer or a smartphone with the internet access at home and
* being able to provide informed consent.

Exclusion Criteria:

* having cognitive, physical, or sensory deficits or language barriers (non-English communicator) that impede study participation
* currently receiving a psychological therapy
* having a prior experience in ACT
* having psychiatric hospitalizations or diagnoses of mental illness in the previous two years
* taking antipsychotic or anticonvulsant medication at the time of recruitment
* considering or planning to place family members of PwD in a nursing home within four months or
* having the possibility of study dropouts due to other medical conditions of family members with dementia (e.g., conditions that may impede study participation due to frequent hospitalization or death)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline to immediately after the intervention and 1 month follow-up on the Depression, Anxiety and Stress Scale | Change from baseline to immediately after the intervention and 1 month follow-up
  Depression, Anxiety and Stress Scale - 21 is a 21-item questionnaire assessing depressive symptoms, anxiety, and stress over the past 7 days on a scale of 0 to 3. Scores on the individual subscales range from 0 to 21. Higher scores indicate greater symptomatology in each subscale of depressive symptoms (7 items), anxiety (7 items), and stress (7 items).
Change from baseline to immediately after the intervention and 1 month follow-up on the Zarit Burden Interview | Change from baseline to immediately after the intervention and 1 month follow-up
  Zarit Burden Interview is a 12-item self-report questionnaire assessing caregiver burden on a scale of 0 to 4. Higher scores indicate higher levels of burden. The total scores range from 0 to 48, and scores of 17 or greater indicate severe/high burden.

SECONDARY OUTCOMES:
Change from baseline to immediately after the intervention and 1 month follow-up on the World Health Organization Quality of Life-BREF - Psychological health component | Change from baseline to immediately after the intervention and 1 month follow-up
  World Health Organization Quality of Life-BREF - Psychological health component has 6 items measuring psychological quality of life. Higher scores denote higher quality of life in terms of psychological health.
Change from baseline to immediately after the intervention and 1 month follow-up on the Meuser Caregiver Grief Inventory | Change from baseline to immediately after the intervention and 1 month follow-up
  Marwit-Meuser Caregiver Grief Inventory Brief-Form is a 6-item self-report questionnaire assessing grief of caregivers. Higher scores indicate higher levels of grief.
Change from baseline to immediately after the intervention and 1 month follow-up on the Caregiver Guilt Questionnaire | Change from baseline to immediately after the intervention and 1 month follow-up
  Caregiver Guilt Questionnaire is a 22-item self-report questionnaire assessing feelings of guilt in caregivers. Higher scores indicate higher levels of guilt.
Change from baseline to immediately after the intervention and 1 month follow-up on the Self-Compassion Scale- Short Form | Change from baseline to immediately after the intervention and 1 month follow-up
  Self-Compassion Scale- Short Form is a 12-item self-report questionnaire assessing self-compassion. Higher scores indicate higher levels of self-compassion.
Change from baseline to immediately after the intervention and 1 month follow-up on the Action and Acceptance Questionnaire-II | Change from baseline to immediately after the intervention and 1 month follow-up
  Action and Acceptance Questionnaire -II is a 7-item self-report questionnaire measuring psychological flexibility. Higher scores indicate poor psychological flexibility.
Change from baseline to immediately after the intervention and 1 month follow-up on the Cognitive Fusion Questionnaire | Change from baseline to immediately after the intervention and 1 month follow-up
  Cognitive Fusion Questionnaire -7 is a 7-item self-report questionnaire measuring cognitive fusion. Higher scores indicate greater levels of cognitive fusion.
Change from baseline to immediately after the intervention and 1 month follow-up on the Engagement in Meaningful Activities Survey | Change from baseline to immediately after the intervention and 1 month follow-up
  Engagement in Meaningful Activities Survey is a 12-item self-assessment instrument that measures a person's subjective experience of the meaningfulness of everyday activities. The total scores range from 12 to 48, and higher scores indicate greater levels of engagement in meaningful activities.

OTHER OUTCOMES:
System Usability Scale | immediately after the intervention
  System Usability Scale (SUS) is a 10-item self-report questionnaire measuring usability of a program/intervention. Higher scores indicate greater levels of perceived usability of the intervention.
Interviews of participants | at baseline and immediately after the intervention
  Caregivers' experiences in the ACT intervention will be explored using individual interviews at posttest. As part of the pretest assessment, we will also explore perceived impacts of COVID-19 on daily lives of family caregivers of people with dementia through individual interviews. Each interview will last for about 30 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Areum Han, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Han A, Yuen HK, Jenkins J. The feasibility and preliminary effects of a pilot randomized controlled trial: Videoconferencing acceptance and commitment therapy in distressed family caregivers of people with dementia. J Health Psychol. 2023 May;28(6):554-567. doi: 10.1177/13591053221141131. Epub 2023 Jan 2. PMID 36591636